CLINICAL TRIAL: NCT00338858
Title: The Connection Between Gait Variability Parameters and Balance Performance in Children With Physical Disability
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alyn Pediatric & Adolescent Rehabilitation Hospital (Other)
Responsible Party: Katz-Leurer, Alyn Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: alyn2CTIL
Record Dates: First submitted 2006-06-19; First posted 2006-06-20 (Estimated); Last update posted 2011-02-15 (Estimated); Status verified 2006-06

CONDITIONS: Brain Injury; Cerebral Palsy
MeSH Terms: conditions — Brain Injuries; Cerebral Palsy | interventions — Walking; Muscle Strength

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Active Comparator): TD
  Interventions: Other: walking and balance performance evaluation; Procedure: muscle strength, walking and balance performance
- 2 (Experimental): TBI
  Interventions: Other: walking and balance performance evaluation; Procedure: muscle strength, walking and balance performance
- a (Experimental): Cerebral palsy
  Interventions: Other: walking and balance performance evaluation; Procedure: muscle strength, walking and balance performance

INTERVENTIONS:
Other: walking and balance performance evaluation
Procedure: muscle strength, walking and balance performance — HHD- muscle strength, Balance performance - TUG, FRT, Walking performance- gaiterite and 2 min walk test

SUMMARY:
The purpose of this study is to explore the connection between gait variability parameters and balance performance in children with physical disability

DETAILED DESCRIPTION:
Step length and step time variability will be measured with an electronic walkway, strength of 4 lower-extremity muscle groups will be tested bilaterally with a hand held dynamometer, walking performance as will be assessed by the 2 minute walk test, energy expenditure index (EEI) and rating of perceived exertion (OMNI scale).

ELIGIBILITY:
Inclusion Criteria:

3 years of age and older Ambulate, with or without an aid

-

Exclusion Criteria:

-

Ages: 3 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2006-06; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hemda Rotem, PT, Principal Investigator — Alyn Hospital
Locations (1):
- Alyn Pediatric and Adolescent Rehabilitation Center, Jerusalem, Israel